CLINICAL TRIAL: NCT06141447
Title: Changes in Rate of Hemorrhage With Prophylactic Oxytocin for Second Trimester Dilation and Evacuation in the Clinic Setting
Brief Title: Changes in Hemorrhage With Prophylactic Oxytocin for Dilation and Evacuation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23-2237
Record Dates: First submitted 2023-11-15; First posted 2023-11-21 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Oxytocin; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial - randomized to either receive treatment (40 units IV oxytocin + 1000 mL normal saline) or placebo (1000 mL normal saline alone).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This will be a double blinded study.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxytocin (Experimental): Participants receive 40 units IV oxytocin in 1000 mL of normal saline at the time of tenaculum placement for D&E.
  Interventions: Drug: Oxytocin + normal saline
- Placebo (Placebo Comparator): Participants receive 1000 mL of normal saline alone at the time of tenaculum placement for D&E.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Oxytocin + normal saline — 40 units IV oxytocin once in a 1000 mL bag of normal saline
  Arms: Oxytocin
Drug: Normal saline — 1000 mL bag of normal saline alone
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness of prophylactic oxytocin on hemorrhage rates for second trimester dilation and evacuation (D&E) in the clinic setting.

ELIGIBILITY:
Inclusion Criteria:

* clinic-based D&E at 18 weeks gestational age and above
* speaks English or Spanish

Exclusion Criteria:

* refuses IV
* history of coagulopathy
* anticoagulant use in the preceding five days
* chorioamnionitis or sepsis
* suspected placenta accreta spectrum
* intrauterine fetal demise
* multiple gestation
* use of misoprostol for cervical preparation

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Hemorrhage | day of procedure
  Quantitative blood loss greater than or equal to 500 mL or a clinical response to excessive bleeding such as transfusion or hospital admission
Quantitative blood loss | day of procedure
  Measured blood loss during procedure

SECONDARY OUTCOMES:
Procedure time | day of procedure
  Length of time of total procedure and length of time until bleeding initially managed

OTHER OUTCOMES:
Patient satisfaction and pain scores | day of procedure
  Patient satisfaction with procedure and maximum reported pain on a visual analog scale
Ease of procedure | day of procedure
  Provider reported ease of procedure
Rate of additional uterotonics | day of procedure
  Report of additional medications to treat bleeding used
Cost of additional uterotonics | day of procedure
  Estimated cost of additional uterotonics used

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Women's Health Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No